CLINICAL TRIAL: NCT06625424
Title: Effect of Short Sprint Interval Training With Active Recovery as Compared to Passive Recovery on Anaerobic Capacity in Non-athletic Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FUI/CTR/2024/38
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Non-athletic Active Young Adults
Keywords: Sprint Interval Training, Non-athletic population young adults, Active Recovery, Passive Recovery, Anaerobic Field Test

STUDY DESIGN:
Intervention Model Description: This study will be a randomized controlled trial (single blinded), consisting of 2 groups: intervention group A (active recovery) and intervention group B (passive recovery).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Participants in this group will perform short sprint interval training on a flat running track in field. Each lane will be materialized by placing cones 5 m from each other for a total of 30 m on which Subject will perform Short Sprint Interval Training.
  The instructions will be to travel the greatest distance possible in 10 seconds, making trips of 5, 10, 15 m, etc.
  Participants of this group will opt for 1 minute of active recovery i.e. they will perform brisk walk between 6 bouts of 10 sec sprint.
  The duration of the training will be of 2 weeks.
  Interventions: Other: Short Sprint Interval Training with Active Recovery
- Control group (Active Comparator): Patients will Participants in this group will perform short sprint interval training on a flat running track in field. Each lane will be materialized by placing cones 5 m from each other for a total of 30 m on which Subject will perform Short Sprint Interval Training.
  The instructions will be to travel the greatest distance possible in 10 seconds, making trips of 5, 10, 15 m, etc.
  Participants of this group will opt for 1 minute of passive recovery i.e. they will stay stationary between 6 bouts of 10 sec sprint.
  The duration of the training will be of 2 weeks.
  Interventions: Other: Short Sprint Interval Training with passive recovery

INTERVENTIONS:
Other: Short Sprint Interval Training with passive recovery — Participants will perform short sprint interval training on a flat running track in field. Each lane will be materialized by placing cones 5 m from each other for a total of 30 m on which Subject will perform Short Sprint Interval Training.
  The instructions will be to travel the greatest distance possible in 10 seconds, making trips of 5, 10, 15 m, etc. Participants will opt for 1 minute of active recovery i.e. they will perform brisk walk between 6 bouts of 10 sec sprint.
  The duration of the training will be of 2 weeks.
  Arms: Control group
Other: Short Sprint Interval Training with Active Recovery — Participants will perform short sprint interval training on a flat running track in field. Each lane will be materialized by placing cones 5 m from each other for a total of 30 m on which the Subjects will perform Short Sprint Interval Training.
  The instructions will be to travel the greatest distance possible in 10 seconds, making trips of 5, 10, 15 m, etc.
  Participants will opt for 1 minute of active recovery i.e. they will perform brisk walk between 6 bouts of 10 sec sprint.
  The duration of the training will be of 2 weeks.
  Arms: Interventional group

SUMMARY:
Short Sprint Interval Training (SSIT) is a modified form of Sprint Interval Training (SIT) defined as "small bouts of supramaximal exercise with recovery periods between them to increase peak oxygen uptake in spite of having a less amount of exercise volume". SSIT was developed so that non- athletic population could also perform a training which was originally designed for athletes to increase anaerobic capacity. The benefit of this type of exercise is that it is time efficient and yields the result in short amount of time as compared to other type of exercises due to its vigorous nature. Moreover this sort of training is mostly performed in lab setting rather than on field, therefore the aim of this study is to determine the effect of short sprint interval training in a field with active recovery as compared to passive recovery on anaerobic capacity in non-athletic population.

DETAILED DESCRIPTION:
Based on a global health initiative to promote "Exercise is Medicine" strategy by American College of Sports Medicine, designing an exercise prescription which is time efficient, cost-effective, easily performable and has great adherence or compliance is necessary. SIT is a type of Anaerobic training which not only enhances the anaerobic capacity but also the aerobic capacity of an individual as well. Thus SIT plays a crucial role in prevention of the NCDs by maintain and improving CRF. Classic SIT is limited to athletic population therefore this study aims to promote the use of modified SIT training protocol called as SSIT by shortening the sprinting time from 30s to 10s so that non-athletic individuals are able to perform it. Apparently there are lack of field based studies on SIT. Most studies use lab based training performed on treadmill and cycle ergometer which can be expensive and time-consuming, especially when several subjects have to train at the same time. Furthermore no comparison has been made between active and passive recovery in short term sprint interval training in field (a bout of 10 second of less). This study aims to test the novel effects of Short Sprint Interval Training with two different types of recovery method performed on field rather than lab to enhance anaerobic capacity in a short amount of time.

This study would be a single blinded randomized control trial, conducted over a period of 12 months at football ground at F-11/1 Islamabad. Subjects will be selected via non-probability convenience sampling technique, followed by block randomization into two groups, the intervention group A and intervention group B using sealed envelope method. The sample size as calculated by G*Power software will be 38 non -athletic individuals. Informed consent will be taken from individuals selected as per inclusion criteria. Participants then being allocated to one of the 2 groups, will be required to complete a self-reporting demographic form. For training, participants will perform SSIT 3 times a week for a total duration of 02 weeks. Anaerobic capacity of the participants will be measured using running based anaerobic sprint test (RAST) before intervention and after intervention of two weeks. Collected data will then be entered and analyzed on the SPSS software version 23.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female young adults ranging from 18-25 Years of age.
* Young adults who perform moderate to vigorous Intensity exercise at least once a week according to IPAQ.
* Those who are cleared for physical activity after screening through PAR-Q.

Exclusion Criteria:

* Young adults having history of any Musculoskeletal, cardiovascular, pulmonary and neurological Disorder.
* Young adults having history of injury in the past 30 days.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Anaerobic Capacity | 2 weeks
  Evaluation will be done using field test known as Running Based Anaerobic Sprint Test (RAST)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan